CLINICAL TRIAL: NCT05020847
Title: The Underlying Causes Affecting the Response to Dietary Rehabilitation in Severely Acutely Malnourished Children at the Center Hôspitalier Universitaire Sourô Sanou, Bobo Dioulasso, Burkina Faso
Brief Title: Effectiveness of Alternative Diets During the Stabilization Phase on Children With Complicated SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); University Hospital Sourô Sanou of Bobo Dioulasso (Burkina Faso) (Unknown); Centre Muraz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-09443-A
Record Dates: First submitted 2021-08-02; First posted 2021-08-25 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Severe Acute Malnutrition; Kwashiorkor; Nutritional Edema; Marasmus
Keywords: Severe acute malnutrition; Nutritional rehabilitation; F75; Stabilization phase; Therapeutic complex of vitamins and minerals (CMV); Kwashiorkor; Marasmus
MeSH Terms: conditions — Severe Acute Malnutrition; Kwashiorkor; Protein-Energy Malnutrition

STUDY DESIGN:
Intervention Model Description: This will be an open, randomized controlled trial aimed at testing the effectiveness of three therapeutic diet regimens during the first phase of hospital management of children with complicated SAM admitted to CREN, Bobo Dioulasso.
  Children aged 6 to 59 months hospitalized in the pediatric department or other services of the Bobo Dioulassso CHUSS, and admitted to the CREN for complicated SAM (WHZ < -3 SD and/or MUAC < 115 mm and/or the presence of nutritional edema) will be randomly assigned to receive:
  1. Standard F75;
  2. Alternative F75 without CMV (mainly containing corn flour, sugar, powdered milk and oil); and
  3. Alternative F75 with CMV (includes most minerals and vitamins like F75 and F100).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard F75 (Active Comparator): At the admission, therapeutic food is given by the nurses every 2 hours on the first day; then if tolerance is good, every 3 hours the following days. No family meals during the stabilization phase. But the baby can breastfeed.
  A child will receive an antibiotic as per the national protocol, malaria treatment if diagnosed with malaria, Vitamin A if symptomatic eye damage, Folic acid in case of anemia, antifungal in case of candidiasis.
  Interventions: Dietary Supplement: Standard F75
- Alternative F75 with CMV (Experimental): At the admission, therapeutic food is given by the nurses every 2 hours on the first day; then if tolerance is good, every 3 hours the following days. No family meals during the stabilization phase. But the baby can breastfeed.
  A child will receive an antibiotic as per the national protocol, malaria treatment if diagnosed with malaria, Vitamin A if symptomatic eye damage, Folic acid in case of anemia, antifungal in case of candidiasis.
  Interventions: Dietary Supplement: Alternative F75 with CMV
- Alternative F75 without CMV (Experimental): At the admission, therapeutic food is given by the nurses every 2 hours on the first day; then if tolerance is good, every 3 hours the following days. No family meals during the stabilization phase. But the baby can breastfeed.
  A child will receive an antibiotic as per the national protocol, malaria treatment if diagnosed with malaria, Vitamin A if symptomatic eye damage, Folic acid in case of anemia, antifungal in case of candidiasis.
  Interventions: Dietary Supplement: Alternative F75 without CMV

INTERVENTIONS:
Dietary Supplement: Standard F75 — F-75 contains 75 kcal and 0.9 g protein per 100 ml
  Arms: Standard F75
Dietary Supplement: Alternative F75 with CMV — Alternative F75 With CMV contains cereal flour, oil, sugar, powdered milk with complex mineral-vitamin (CMV)
  Arms: Alternative F75 with CMV
Dietary Supplement: Alternative F75 without CMV — Alternative F75 without CMV contains cereal flour, oil, sugar, powdered milk without complex mineral vitamin (CMV).
  Arms: Alternative F75 without CMV

SUMMARY:
Severe acute malnutrition (SAM) is a life threatening condition and is defined by 1) a weight-for-height Z-score more than three standard deviations (SD) below the median based on the 2006 World Health Organization (WHO) growth standards, 2) a mid-upper arm circumference (MUAC) of less than 115 mm or 3) by the presence of nutritional edema. Signs such as edema, mucocutaneous changes, hepatomegaly, lethargy, anorexia, anemia, severe immune deficiency and rapid progression to mortality characterize a state commonly coined as "complicated SAM". Kwashiorkor is one of the forms of complicated SAM commonly distinguished by the unmistakable presence of bipedal edema. SAM results in high mortality rates of up to half a million child deaths annually. Undernourished children are at higher risk of mortality ranging from three times more risk among children with moderate malnutrition to 10-times in SAM children compared to well-nourished children. Children with complicated SAM require inpatient treatment in specialized centers.

The "Rehabilitation and Nutritional Education Center" (CREN) is a specialized center in Burkina Faso receiving on average 10 SAM children per day. Recovery rate is lower than international standards; and adverse events and mortality remain strikingly high.

Our main objective is to assess the underlying risk factors affecting the effectiveness of the nutritional therapeutic treatment protocol for complicated SAM children under 5 years of age who have been referred to the CREN, at the Centre Hôspitalier Universitaire Souro, Bobo Dioulasso, Burkina Faso.

The specific objective is to assess the effectiveness of alternative dietary regimens during the stabilization phase on well-specified clinical and biochemical outcomes in children with complicated SAM. Dietary regimens differ by their carbohydrate profile and content, and by their different micronutrient composition including vitamin A, iron and zinc.

DETAILED DESCRIPTION:
Severe acute malnutrition (SAM), defined as severe wasting [weight-to-height Z-score < -3 standard deviations (SD), based on the WHO Child Growth Standards] and / or the presence of nutritional edema, and / or mid-upper arm circumference (MUAC) <115 mm, is a condition that requires urgent attention and appropriate management to reduce mortality and promote recovery among children. Management of SAM children without complications is provided at the community level. Hospitalization in specialized care centers is necessary for SAM children with complications. SAM children with comorbidities have a greater risk of mortality and treatment failure. Our knowledge of the specific adequate nutritional needs of SAM is limited.

For the treatment of SAM in hospital, the WHO recommends the use of therapeutic milk low in protein 'F75' in the stabilization phase; and more protein-rich F100 or F75 combined with ready-to-use therapeutic foods (RUTF) in the transition phase. The WHO also recommends using as an alternative formula made of cereal flour, skimmed milk powder, oil, sugar, and a therapeutic vitamin and mineral complex (CMV), in case of shortage of the standard therapeutic milk F75 / F100 or in case of signs of intolerance (vomiting, diarrhea).

The Refeeding Center - Centre de Récupération et d'Education Nutritionnelle (CREN) of the Sourô Sanou University Hospital Center (CHUSS) in Burkina Faso specializes in the care of SAM children with complications. In 2018, out of 500 children aged 6-59 months admitted for SAM with complications, the CHUSS CREN registered 86.8% full recovery, 8.2% dropout and 5% death. Although the recovery rate is higher than international standards (greater than 75%), the mortality rate remains higher than the recommended 3% by international standards; in addition to the challenges that are faced locally in maintaining high standards of care. At the CREN, we observed that some SAM children with complications can have severe diarrhea and vomiting after taking F75 (first phase of the nutritional treatment). It was also observed that other SAM children with edema, whose edema resolved in the first phase of treatment under F75, redeveloped edema when they received RUTF (Plumpy Nut®) in the transition phase according to the WHO 2013 protocol.

The second objective of the study is to assess the risk factors affecting the response to dietary treatment in this center (the CREN, Burkina Faso) and to compare alternatives for treatment during the nutritional rehabilitation.

Problematic It was observed at the Refeeding Center (CREN) of the Sourô Sanou University Hospital (CHUSS) in Bobo Dioulasso, that SAM children with complications show during their treatment, signs of intolerance to F75 (diarrhea , vomiting). The pathophysiology of diarrhea in SAM involves several theories including that of lactose intolerance, and that of alteration of the intestinal microbiota.

The study aims to assess the effectiveness of diet regimens [standard F75, or alternative F75 + mineral vitamin complex (CMV), or alternative F75 without CMV] during the stabilization phase from both a clinical and biochemical aspects in children with complicated SAM. Diets differ in their profile and carbohydrate content, and in their different micronutrient compositions, including vitamin A, iron and zinc.

Our hypothesis is that the F75 alternative during the stabilization phase (the first phase) of complicated SAM children is associated with better compliance, less diarrhea and better outcomes than the recommended F75 formulation; and that children treated correctly with the F75 alternative containing CMV will perform better than the other two groups of children treated with F75 or the F75 alternative without CMV.

This will be an open, randomized controlled trial aimed at testing the effectiveness of three therapeutic diet regimens during the first phase of hospital management of children with complicated SAM admitted to CREN, Bobo Dioulasso.

After obtaining informed consent from parents / guardians for the inclusion of the child, the child will be randomized and will receive their assigned treatment. In accordance with the 2014 protocol for the management of SAM in Burkina Faso, an antibiotic will be given as part of the systematic treatment of complicated SAM, and other medical treatments depending on the associated complication. Deworming is provided also gratis, will be done only in children whose tests are positive for intestinal parasites and ONLY in the rehabilitation phase (the third phase of the treatment) as per the National Protocol for the management of complicated SAM. The dietetic treatment will be given by the nurses every 2 hours on the first day; then if tolerance is good, every 3 hours the following days. No family meals during phase 1. But the baby can breastfeed. The observance and tolerance of the treatment will be noted by the nurses: amount of milk taken, refusal, vomiting, diarrhea, presence of a nasogastric tube. The quantities will be given according to the weight of the child, the presence or not of edema, in accordance with the national protocol.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute malnutrition defined as Weight-for-Height Z-score (WHZ) <- 3 SD AND / OR MUAC <115 mm AND / OR with edema
* With complications
* Who are admitted and treated in the refeeding center (CREN) of the CHUSS
* Aged between 6 and 59 Months
* Parental Signed informed consent form

Exclusion Criteria:

* Children younger than 6 months or older than 59 months of age
* Moderate Acute Malnutrition (MAM)

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Recovery rate of children | Three to Five days
  Number of children treated and admitted to the transition phase
Daily weight gain | Three to Five days
  Average daily weight gain in the stabilization phase in Grams
Number of days during the first phase of treatment | Three to Five days
  Average number of days spent in the stabilization phase in Day

SECONDARY OUTCOMES:
% of intake of the therapeutic regimen | Three to Five days
  Daily intake of the administered dietary treatment
Anorexia | Three to Five days
  Serious severe event that occurs at anytime during the treatment
Mortality | Three to Five days
  Serious severe event that occurs at anytime during the treatment
Diarrhea | Three to Five days
  Serious severe event that occurs at anytime during the treatment
Vomiting | Three to Five days
  Serious severe event that occurs at anytime during the treatment

OTHER OUTCOMES:
HIV/AIDS | Three to Five days
  Detection of HIV/AIDS using polymerase chain reaction (PCR) in infants and children younger than 18 months or retroviral serology test in older children.
Hepatitis infection | Three to Five days
  Blood test of hepatitis using the enzyme-linked immunosorbent assay (ELISA)
Tuberculosis infection | Three to Five days
  Test of tuberculosis via search for Koch's Bacillus in gastric/spit tubing and molecular testing of stools using polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — University Ghent; Jerome Some, Md. PhD, Principal Investigator — Institut de Recherche en Sciences de la Sante, Burkina Faso; Bintou Sanogo, MSc. Md., Principal Investigator — Centre Hospitalier Universitaire Souro, Bobo Dioulasso, Burkina Faso.
Locations (1):
- Centre Hospitalier Universitaire Souro, Bobo-Dioulasso, Bobo Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: No
All the data that can affect the main or the secondary outcomes will be used in the analyses and shared as necessary.

REFERENCES:
- [Background] Singh K, Badgaiyan N, Ranjan A, Dixit HO, Kaushik A, Kushwaha KP, Aguayo VM. Management of children with severe acute malnutrition: experience of Nutrition Rehabilitation Centers in Uttar Pradesh, India. Indian Pediatr. 2014 Jan;51(1):21-5. doi: 10.1007/s13312-014-0328-9. Epub 2013 Jul 5. PMID 24277964
- [Background] Nguefack F, Adjahoung CA, Keugoung B, Kamgaing N, Dongmo R. [Hospital management of severe acute malnutrition in children with F-75 and F-100 alternative local preparations: results and challenges]. Pan Afr Med J. 2015 Aug 31;21:329. doi: 10.11604/pamj.2015.21.329.6632. eCollection 2015. French. PMID 26587175
- [Background] Gopalan C. Kwashiorkor and marasmus: evolution and distinguishing features. 1968. Natl Med J India. 1992 May-Jun;5(3):145-51. No abstract available. PMID 1306670
- [Background] Bartz S, Mody A, Hornik C, Bain J, Muehlbauer M, Kiyimba T, Kiboneka E, Stevens R, Bartlett J, St Peter JV, Newgard CB, Freemark M. Severe acute malnutrition in childhood: hormonal and metabolic status at presentation, response to treatment, and predictors of mortality. J Clin Endocrinol Metab. 2014 Jun;99(6):2128-37. doi: 10.1210/jc.2013-4018. Epub 2014 Feb 27. PMID 24606092
- [Background] Deen JL, Funk M, Guevara VC, Saloojee H, Doe JY, Palmer A, Weber MW. Implementation of WHO guidelines on management of severe malnutrition in hospitals in Africa. Bull World Health Organ. 2003;81(4):237-43. Epub 2003 May 16. PMID 12764489
- See also: World Health Organization (2013) WHO guideline: updates on the management of severe acute malnutrition in infants and children. — https://www.who.int/publications/i/item/9789241506328
- See also: Enquête Nutritionnelle Nationale SMART 2016 au Burkina Faso. 2016 ; 47p — https://www.unicef.fr/article/malnutrition-la-situation-au-burkina-faso
- See also: Ministère de la Sante au Burkina Faso. Protocol National : Prise en charge intégrée de la malnutrition aigüe (PCIMA). 2014 — https://www.humanitarianresponse.info/sites/www.humanitarianresponse.info/files/documents/files/protocole_pcima_bf_janv_2015.pdf